CLINICAL TRIAL: NCT00728026
Title: Autonomic Profiles in Pediatric Patients With Cyclic Vomiting Syndrome, Irritable Bowel Syndrome, Postural Orthostatic Tachycardia Syndrome, Functional Abdominal Pain or Chronic Nausea
Brief Title: Autonomic Profiles in Pediatric Patients With Cyclic Vomiting Syndrome (CVS), Irritable Bowel Syndrome (IBS),Postural Orthostatic Tachycardia Syndrome (POTS), Functional Abdominal Pain (FAP) or Chronic Nausea
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, B Li, Professor of Pediatrics, Medical College of Wisconsin
Other Study IDs: 08/112; GC 680
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Vomiting Syndrome; Irritable Bowel Syndrome; Postural Orthostatic Tachycardia Syndrome; Abdominal Pain; Chronic Nausea
Keywords: Chart must reveal the following procedures:; Heart rate variability,; Deep Breathing Test,; Valsalva maneuver,; Table test,; Thermoregulatory Sweat Testing,; Quantitative Sudomotor Axon Reflex Test (QSART),; Vital signs,; postural changes in heart rate and blood pressure,; composite autonomic score
MeSH Terms: conditions — Irritable Bowel Syndrome; Postural Orthostatic Tachycardia Syndrome; Abdominal Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Cyclic Vomiting Syndrome
- 2: Irritable Bowel Syndrome
- 3: Postural Orthostatic Tachycardia Syndrome
- 4: Functional Abdominal Pain
- 5: Chronic Nausea

SUMMARY:
Retrospectively review the charts of all children who had heart rate variability, deep breathing test, valsalva maneuver, tilt table test, thermoregulatory sweat testing, quantitative sudomotor axon reflex test (QSART) completed and were cared for at Children's Hospital of Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient services

Exclusion Criteria:

* Inpatient services

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of either: Cyclic Vomiting Syndrome (CVS), Irritable Bowel Syndrome (IBS), Chronic nausea, Postural Orthostatic Tachycardia Syndrome (POTS), Functional Abdominal Pain (FAP)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2008-06; Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
To gather preliminary data to characterize autonomic function in children and adolescents with functional gastrointestinal disorders. | One year

CONTACTS AND LOCATIONS:
Overall Officials: B UK Li, Principal Investigator — Medical College of Wiconsin